CLINICAL TRIAL: NCT05289804
Title: Diminishing Accelerated Long-term Forgetting in Mild Cognitive Impairment: Study Protocol for a Prospective, Double-blind, Placebo-controlled, Randomized Controlled Trial
Brief Title: Diminishing Accelerated Long-term Forgetting in Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPREC102021-23; AARG-21-848486 (Other Grant/Funding Number: Alzheimer's Association Research Grant)
Record Dates: First submitted 2022-02-22; First posted 2022-03-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Memory Impairment; Memory Disorders in Old Age
Keywords: episodic memory; amnestic mild cognitive impairment; mild Alzheimer's disease; electrical stimulation; greater occipital nerve
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders | interventions — Transcutaneous Electric Nerve Stimulation; Lidocaine; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: The investigators have opted to use a parallel-group design as it is unclear what the carry-over effect and/or wash-out period will be for NITESGON. Patients will be randomized after the baseline evaluation and will be assigned to receive one of the four possible types of NITESGON. To eliminate subjective bias, all patients and the investigator testing the endpoint measures will be blinded to the type of intervention.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active NITESGON (Experimental): One electrode each will be placed over the left and right C2 dermatomes. A constant current will be applied during the word association task.
  Interventions: Device: NITESGON
- Sham NITESGON (Sham Comparator): For sham NITESGON (inactive control), placement of the electrodes will be identical to active NITESGON. Current intensity (ramp down) will gradually be reduced as soon as NITESGON reaches a current flow of 1.5 mA. The rationale behind this sham procedure is to mimic the transient skin sensation at the beginning of active NITESGON without producing any conditioning effects on the brain.
  Interventions: Device: Sham NITESGON
- Active NITESGON + local anesthesia (Active Comparator): For active NITESGON + local anesthesia (active control; local nerve anesthesia group), patients will receive NITESGON, in combination with a topical skin anesthetic (lidocaine/prilocaine cream) to reduce any potential contribution from transcutaneous stimulation of peripheral nerves. A current similar to active NITESGON will be applied.
  Interventions: Device: NITESGON; Drug: Lidocaine / Prilocaine Topical Cream
- Active C5/C6 (Active Comparator): For the active C5/C6 group (active control; same sensation different nerve), the electrodes will be placed over cervical nerves five and six, to mimic the sensation, but change the location. A current similar to active NITESGON will be applied.
  Interventions: Device: C5/C6 stimulation

INTERVENTIONS:
Device: NITESGON — NITESGON will be delivered by a specially developed, battery-driven, constant current stimulator via a pair of saline-soaked surface sponges on the scalp. One electrode each will be placed over the left and right C2 dermatomes.
  NITESGON will first be switched on in a ramp-up fashion over 30 seconds. For active NITESGON, stimulation will occur during the word association task. For sham the current intensity (ramp down) will gradually be reduced (over 5 seconds) as soon as NITESGON reaches a current flow of 1.5 mA. The rationale behind this sham procedure is to mimic the transient skin sensation at the beginning of active NITESGON without producing any conditioning effects on the brain.
  Other Names: non-invasive transcutaneous electrical stimulation of the greater occipital nerve; transcutaneous electrical stimulation; tES; stimulation
  Arms: Active NITESGON; Active NITESGON + local anesthesia
Drug: Lidocaine / Prilocaine Topical Cream — A topical skin anesthetic (lidocaine/prilocaine cream) will be used to reduce any potential contribution from transcutaneous stimulation of peripheral nerves. This lidocaine/prilocaine preparation blocks sodium channels in peripheral nerves in the skin and thereby stabilizes the membrane potential and increases the threshold for firing an action potential.
  Other Names: lidocaine/prilocaine cream; local anesthetic
  Arms: Active NITESGON + local anesthesia
Device: C5/C6 stimulation — The electrodes will be placed over cervical nerves five and six, to mimic the sensation, but change the location.
  Arms: Active C5/C6
Device: Sham NITESGON — Sham NITESGON
  Arms: Sham NITESGON

SUMMARY:
This study is designed as a prospective, double-blind, placebo-controlled, randomized parallel-group study that will be completed at the clinical research facility at St. James' Hospital and at Trinity College Dublin, Ireland. A total of 100 amnestic mild cognitive impairment (aMCI) patients will receive a (real or control) non-invasive transcutaneous electrical stimulation procedure. Patients will be assigned to one of four groups. One group will receive active stimulation, while the three groups will be control groups. One groups will be receive sham stimulation (inactive control), while a second group will receive active stimulation and local anesthesia and a third group will stimulate a different nerve (active control; same sensation different nerve). The investigators will include three control groups to verify that the effect is real and location specific and cannot be associated to a sensation effect. The investigators have opted to use a parallel-group design as it is unclear what the carry-over effect and/or wash-out period will be for stimulation. To eliminate subjective bias, all patients and the investigator testing the endpoint measures will be blinded to the type of intervention. The primary outcome, i.e. memory recall, will be determined by a word association task recorded immediately after stimulation, 7 days after stimulation, and 28 days after stimulation. The secondary outcomes is neurophysiological changes determined by resting state EEG, which will be assessed immediately before and after stimulation in the first session.

The investigators will conduct this study as follows:

1. Screening aMCI patients.
2. Randomly assigning aMCI patients to one of the four groups.
3. Administering one session active stimulation (n = 25) or control (n = 25 in each of three control group) stimulation paired with a word-association task; administered by research assistant.
4. Behavioral assessments after each of the three blocks of studying the word associations and neural measures immediately after the last session of Behavioral assessments (T0).
5. Behavioral assessments at seven (T1) and 28 (T2) days after stimulation.

DETAILED DESCRIPTION:
Patients 50 years of age and above with amnestic mild cognitive impairment (aMCI), will be recruited to the memory clinic at St. James and the Memory Assessment and Support Service Tallaght University Hospital. The investigators plan to include 100 English-speaking aMCI patients. To participate in this study, subjects should be able to provide an informed consent, have a confirmed aMCI diagnosis and have their medication stable for at least three months prior to baseline data collection. Prospective participants, who meet the criteria, will be sent an electronic copy of the consent form. Participants will only be asked to sign the consent form at the site after going over the form with the researcher where all aspects of the study protocol will be reviewed.

The study is designed to give us adequate power to detect clinically meaningful differences between the groups. Twenty individuals per group (total n = 80) would offer us a power of 80% to detect the difference between groups using Cohen's d estimation of effect size. A sample size of 80 will allow us to see a large effect size. Although The investigators do not expect attrition to be large, a dropout rate of no more than 10% is expected. This trial is longitudinal which could increase its drop-out rate. The investigators will thus oversample to a target sample size of 25 patients per group to assure that our power to detect effects is maintained. The overall sample will be 100. The investigators aim to recruit patients with aMCI and display pre-symptomatic signs of Alzheimer's disease (AD). An age ranging from 50 years and above is a good fit for this population.

The study consists of three in person sessions. Session 1 will consist of a word association memory task in which participants are instructed to memorize a subset of words. Participants will either receive active stimulation or control stimulation during the word-association task. Session 1 will also include demographic and mood related questionnaires, as well as EEG before and after memory testing. At the end of EEG testing, participants will fill out an exit questionnaire developed by Brunoni et al. to assess potential side-effects (headache, neck pain, scalp pain, tingling, itching, burning sensation, skin redness, sleepiness, trouble concentrating, mood changes) at the end of stimulation. One week after Session 1, Session 2 will take place. They will again complete the word association memory task. Three weeks after Session 2, Session 3 will take place and participants will complete the word association memory task and complete a blinding questionnaire at the end of the session.

During memory testing, participants will receive one of four interventions. Participants will encounter a second researcher who will take over for the first researcher in order to provide the blinded-stimulation protocol. They will be assigned randomly (like a flip of a coin) to one of four groups. Some groups will receive active stimulation and the other three groups will serve as controls. For sham stimulation, placement of the electrodes will be identical to active stimulation. A third group will receive stimulation, but with a topical skin anesthetic. For the fourth control group, the electrodes will be placed on the lower neck. For both the third and fourth control group, the current similar to active stimulation will be applied.

Participants will be paid at the end of the session and will be asked to sign a receipt of the money. If they successfully complete the study, they will be compensated for travel with 10 euros, if they wish to withdraw or are unable to proceed because of any in-eligibility in the in-person session, they will be compensated with 5 euros for travel.

All data will be managed using unique study codes, which will be used to code and file all electronic information, to protect participant confidentiality. To ensure privacy, all research files (e.g. screening, consent, questionnaires) will be stored in locked file cabinets in locked offices at Trinity. Electronic information (e.g. EEG and behavioral data) will be stored at a secure, password-protected, server at Trinity and all corresponding data analysis will be conducted at Trinity to ensure central and complete data protection. Subject names will not be published. Summary statistics will be performed on all variables and reported. The person processing the data will not be able to trace back the data to the individual. Data will contain a pseudonymised subject code and thus be de-identified. Pseudonymised data will be stored for 7 years as required by GDPR rules. After this personal and raw data will be deleted and the data will be anonymised. The processed data and group analysis will stored be indefinitely and will be shared through Trinity TARA Open Access database to promote Open Science. The key codes linking the participant names to the pseudonymised data will be stored in a secure Excel file in a secure USB by the Principal Investigator.

An intention-to-treat and per-protocol analysis will be performed. For the intention-to-treat analysis, the patient must successfully complete T0 and T1 assessments. For missing observations, the Last Observation Carried Forward (LOCF) approach will be used. Exclusion from the population will be finalized prior to database lock in a blinded manner. Memory recall during the word-association task will be assessed to determine memory performance. For EEG data, sLORETA statistical contrast maps will be calculated for the sham and active groups through multiple voxel-by-voxel comparisons in a logarithm of F-ratio. For transcutaneous electrical stimulation (TES) adverse events, a comparison will be conducted between the active and sham group using a one-way ANOVA with stimulation (active vs sham) as independent variable and adverse events as dependent variable. A Chi-square test will be conducted comparing actual stimulation (active vs sham) versus participants' expected stimulation (active vs sham) to determine if subjects were blinded to the experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years
* Diagnosis of probable aMCI or mild AD
* Montreal Cognitive Assessment between 18-25
* Mini Mental State Examination score >21
* Stable AChl medication >3 months
* Adequate visual and auditory acuity
* Capacity to understand and sign informed consent

Exclusion Criteria:

* Any cause of cognitive decline or dementia that is not Alzheimer's disease related including parkinsonism related dementias, vascular dementia, fronto-temporal dementia.
* Enrolment in an ongoing investigational medicinal product study
* History in the past 2 years of epileptic seizures
* Any current major psychiatric disorder
* Evidence of brain damage, including significant trauma, stroke, hydrocephalus, intellectual disability, or serious neurological disorder.
* History of alcoholism or drug abuse within the last 12 months
* Medical devices not eligible for MRI scanning

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Word association task performance immediately after NITEGON/sham | Patients will be tested immediately after NITESGON/sham (T0)
  Patients will perform a Swahili-English word association task. Patients will be asked to learn a list of 50 Swahili-English word pairs. In a test phase, patients will be presented with the Swahili word and asked to type the correct English translation.
Word association task performance at 7 days | 7 days after NITESGON/sham (T1)
  Patients will be asked to return for a follow-up test 7 days later. The test will be identical to the test phase from T0 timepoint.
Word association task performance at 28 days | 28 days after NITESGON/sham (T2)
  Patients will be asked to return for a follow-up test 28 days after NITESGON/sham. The test will be identical to the test phase from T0 timepoint.

SECONDARY OUTCOMES:
EEG gamma oscillations | Resting state EEG will be collected immediately before and immediately after NITESGON/sham.
  Rest-state EEG will be collected immediately before and after NITESGON/sham (T0) and will be correlated with the recall of the word-association task 7 (T1) and 28 (T2) days after NITESGON.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- TCIN, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Luckey AM, McLeod SL, Robertson IH, To WT, Vanneste S. Greater Occipital Nerve Stimulation Boosts Associative Memory in Older Individuals: A Randomized Trial. Neurorehabil Neural Repair. 2020 Nov;34(11):1020-1029. doi: 10.1177/1545968320943573. Epub 2020 Sep 23. PMID 32964776
- [Background] Vanneste S, Mohan A, Yoo HB, Huang Y, Luckey AM, McLeod SL, Tabet MN, Souza RR, McIntyre CK, Chapman S, Robertson IH, To WT. The peripheral effect of direct current stimulation on brain circuits involving memory. Sci Adv. 2020 Nov 4;6(45):eaax9538. doi: 10.1126/sciadv.aax9538. Print 2020 Nov. PMID 33148657
- [Derived] Adcock KS, Lawlor B, Robertson IH, Vanneste S. Diminishing accelerated long-term forgetting in mild cognitive impairment: Study protocol for a prospective, double-blind, placebo-controlled, randomized controlled trial. Contemp Clin Trials Commun. 2022 Sep 2;30:100989. doi: 10.1016/j.conctc.2022.100989. eCollection 2022 Dec. PMID 36117569